CLINICAL TRIAL: NCT01457144
Title: First Line Mantle Cell Lymphoma (MCL) Treatment by RiBVD Schema in Patients Older Than 65 Years or 18 to 65 Years Old Who Cannot or Refuse Receive Conditioning Regimen Followed by Autograft
Brief Title: Study of Mantle Cell Lymphoma Treatment by RiBVD
Acronym: RIBVD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Lymphoma Study Association (Other); Janssen-Cilag Ltd. (Industry); Mundipharma Pte Ltd. (Industry); Roche Pharma AG (Industry); Chugai Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Manteau RiBVD
Record Dates: First submitted 2011-10-20; First posted 2011-10-21 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Rituximab; bendamustine; Velcade; Dexamethasone
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RiBVD (Experimental): Rituximab Bendamustine Velcade® Dexamethasone 6 cycles every 28 days
  Interventions: Drug: RiBVD

INTERVENTIONS:
Drug: RiBVD — Every cycle:
  Rituximab intravenous infusion dosage 375 mg/m² day 1 Bendamustine direct intervenous 90 mg/m² day 1 and day 2 Velcade®subcutaneous 1,3 mg/m² day 1,4, 8 and 11 dexamethasone 40 mg IVD on day 2

SUMMARY:
Study of First line mantle cell lymphoma treatment by Rituximab, Velcade, Bendamustine and Dexamethasone schema in patients older than 65 years or 18 to 65 years old who cannot or refuse receive conditioning regimen followed by autograft.

DETAILED DESCRIPTION:
Demonstration of Improvement of progression-free survival (PFS) compared to literature data. 6 months prolongation equal 24 months compared to 18 months obtained whatever the current regimen and in particular compared to RCHOP regimen

ELIGIBILITY:
Inclusion Criteria:

* mantle cell Lymphoma CD20 positive
* Untreated patients
* 65 ans years old patients or 18 to 65 years old patients who can't or refuse receive conditioning regimen followed by autograft.
* Stages Ann Arbor II, III or IV,
* ECOG performance status of 0, 1 or 2
* Without history of neoplasm, except in situ cervix carcinoma and cutaneous basal cell epithelioma, or in complete remission since 3 years,
* Without drug contraindication used in the schema (Rituximab, benda-mustine, Velcade, Dexamethasone),
* Without heart insufficiency or stabilized,
* With the following biological values limits except if pathological values are due to Medullary invading or hypersplenism, hepatic involvement) :PNN more than 1 G/L, Platelets more than 50 G/L,Transaminases (SGOT and SGPT) and alkalin phosphatases alcalines less than 4 x normal,Bilirubin less than 3 x N,- Clearance creatinemia more than 20 mL/min
* Hepatitis B negative serology unless the seropositivity is clearly linked to a vaccination.
* Can be regularly followed
* Who signed the informed consent,
* Affiliated to a national insurance or such a same scheme .

Exclusion Criteria:

* Other type of lymphoma than mantle cell lymphoma according to OMS 2008 classification
* Patients in relapse, except those in relapse due to localized stade who only received locoregional irradiation or splenectomized,
* Central nervous system localization in particular meninge,
* Drug used in the schema contraindication Rituximab , Bendamustine , Velcade® or Dexamethasone
* Non stable diabetes,
* HIV positive or active hepatitis C or B
* ECOG performance status equal or more than 3
* Peripheral neuropathy, whatever its origin, rated more than 2 from NCI
* Non stabilized heart insufficiency,
* Patient who can't receive hyperhydration in order to treat tumoral lysis syndrome or in prophylaxis,
* Patient who can't, whatever the reason, be regularly followed,
* Major patient who are on legal protection, or can't give their consent
* Patient who has not signed the informed consent

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Improvement of progression-free survival (PFS) | 18 months
  Improvement of progression-free survival (PFS) compared to litterature data 6 months prolongation 24 months compared to 18 months obtained whatever the current regimen and in particular compared to RCHOP regimen in reference with Lenz JCO 2005

SECONDARY OUTCOMES:
Overall and complete response rate after 4 cures and 6 cures | 6 months
  Overall and complete response rate after 4 cures equal intermediate response and after 6 cures equal final response according to Cheson 1999 criteria without Positron Emission Tomography and 2007 with Positron Emission Tomography
Residual disease evaluated by molecular biology | 6 years
  Residual disease evaluated by molecular biology on blood and bone marrow, by Hybridation Fluorescente In Situ and Flow cytometry on blood cells
Intermediate response predictive factors study | 4 months
  Predictive factors are determined at diagnosis are watched at Intermediate response
Toxicity of RiBVD regimen according to NCI criteria Hematological and non-hematological toxicity | 6 months
  Toxicities are collected at every course = every 28 days during 6 months
Prognosis value on Overall survival and progression free survival and on duration of response, of the MIPI index, MIPIb index and goelams index | 36 months
Residual disease evaluated by molecular biology Q-PCR on blood and bone marrow, by Hybridation Fluorescente In Situ and Flow cytometry on blood cells | 42 months
  blood and bone marrow samples sent to central laboratory for molecular residual disease at diagnosis, treatment evaluation and follow-up
Diagnostic PET scan results, at intermediate and final analysis | 4 and 6 months
  Pet scan results at intermediate analysis = 4 months Pet scan results at final analysis = 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rémy GRESSIN, MD, Principal Investigator — Groupe Est Ouest des Leucémies et autres Maladies du Sand
Locations (1):
- Valerie ROLLAND NEYRET, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FILO internet site — http://www.filo-leucemie.org